CLINICAL TRIAL: NCT05584826
Title: MDMA-assisted Therapy for Adjustment Disorder (AD) in Dyads of Patients With Cancer and a Concerned Significant Other
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunstone Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSAD1
Record Dates: First submitted 2022-10-10; First posted 2022-10-18 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Adjustment Disorders
MeSH Terms: conditions — Neoplasms; Adjustment Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDMA-Assisted Therapy (Experimental): Participants will receive two doses of MDMA, administered during the Treatment Period with manualized therapy. This 8-week Treatment Period includes two Preparatory Sessions and four Integrative Sessions of non-drug therapy.
  Interventions: Drug: MDMA

INTERVENTIONS:
Drug: MDMA — On 2 separate treatment visits, participants will receive dosing of 100 mg MDMA HCl (~84 mg MDMA) + 40 mg MDMA HCl (~34 mg MDMA) supplement unless tolerability issues arise from the first dose or the participant declines
  Other Names: 3,4-methylenedioxymethamphetamine (MDMA)

SUMMARY:
The goal of this clinical trial is to assess feasibility, tolerability and preliminary effectiveness of MDMA-assisted therapy for adjustment disorder (AD) in 10 dyads of patients with cancer and a concerned significant other (CSO) (20 participants total).

Participants will undergo an 8-week treatment period which will include two doses of MDMA, two Preparatory Sessions and four Integrative Sessions of non-drug therapy.

DETAILED DESCRIPTION:
This open-label single site concurrent mixed-method phase 2 pilot trial will assess the feasibility, tolerability and preliminary effectiveness of MDMA-assisted therapy for adjustment disorder (AD) in 10 dyads of patients with cancer and a concerned significant other (CSO) (20 participants total). The intervention will include two doses of MDMA, administered during the Treatment Period with manualized therapy. This 8-week Treatment Period includes two Preparatory Sessions and four Integrative Sessions of non-drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years old
2. Are considered important to their well-being by patient participants (e.g., spouse or close family member)
3. Meet DSM-5 criteria for current AD (no criteria for another mental disorder and does not correspond to an exacerbation of a preexisting mental disorder. Does not represent a normal bereavement)
4. Satisfies diagnostic criteria for AD using the ADNM-2020 (score ≥ 47.5 on the scale)
5. Are able to swallow pills.
6. Are willing to be driven home after the experimental sessions, either by a driver arranged by the participant or by the site personnel or taxi and agree not to drive after each Experimental Session until the therapists deem it safe to do so
7. If able to become pregnant (i.e. assigned female at birth, fertile, following menarche and until becoming post-menopausal unless permanently sterile), must have a highly sensitive negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session. Adequate birth control methods include intrauterine device (IUD), injected, implanted, intravaginal, or transdermal hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner, or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e. condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom).
8. Must agree to inform the Clinical Investigators within 48 hours of any medical conditions and procedures
9. Are proficient in speaking and reading English
10. Agree to have all clinic visit sessions recorded to audio and video
11. Agree to the following lifestyle modifications (described in more detail in Section 4.3 Lifestyle Modifications): comply with requirements for fasting and refraining from certain medications prior to Experimental Sessions, not enroll in any other interventional clinical trials during the duration of the study, be driven home after each Experimental Session, and commit to medication dosing, therapy, and study procedures.
12. May have well-controlled hypertension that has been successfully treated with anti-hypertensive medicines, if they pass additional screening to rule out underlying cardiovascular disease.
13. May have asymptomatic Hepatitis C virus (HCV) that has previously undergone evaluation and treatment as needed.
14. May have alcohol or substance use disorder if participant is not in withdrawal or requiring detox. Participants must have a plan, agreed upon by investigator, therapy team, and study physician, to reduce use of alcohol or other substances and to manage symptoms without self-medicating. Enrollment will require that, in the judgment of the investigator, therapy team, and study physician, the plan for decreasing substance use is realistic and has a good chance of succeeding in order to prevent substance use from impacting the safety or efficacy of the investigational treatment.
15. May have a history of or current Diabetes Mellitus (Type 2) if additional screening measures rule out underlying cardiovascular disease, if the condition is judged to be stable on effective management, and with approval by the study physician.
16. May have hypothyroidism if taking adequate and stable thyroid replacement medication.
17. May have a history of, or current, glaucoma if approval for study participation is received from an ophthalmologist.

Exclusion Criteria:

1. Concurrent or recent (less than four weeks) cytotoxic chemotherapy or radiation therapy, that impairs general level of physical functioning (index participant)
2. Weigh less than 48 kg
3. Condition impairing oral intake or digestive absorption
4. Are not able to give adequate informed consent
5. Significant suicide risk as defined by suicidal ideation with intend and a plan as endorsed on items 5 on the C-SSRS within the past 6 months or at V0 (see Appendix A)
6. Have any current problem which, in the opinion of the investigator or study physician, might interfere with participation
7. Would present a serious risk to others as established through clinical interview and contact with treating psychiatrist.
8. Have a history of, or a current primary psychotic disorder, major depressive disorder with psychotic features, bipolar affective disorder type 1 or history of or current dissociative identity disorder
9. Require ongoing concomitant therapy with a psychiatric medication with exceptions described in Section 8.0: Concomitant Medications.
10. Have received Electroconvulsive Therapy (ECT) within 12 weeks of enrollment.
11. Have used Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the first Experimental Session;
12. Have a history of ventricular arrhythmia at any time, other than occasional premature ventricular contractions (PVCs) in the absence of ischemic heart disease.
13. Have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation.
14. Have a history of arrhythmia, other than premature atrial contractions (PACs) or occasional PVCs in the absence of ischemic heart disease, within 12 months of screening.

    Participants with a history of atrial fibrillation, atrial tachycardia, atrial flutter or paroxysmal supraventricular tachycardia or any other arrhythmia associated with a bypass tract may be enrolled only if they have been successfully treated with ablation and have not had recurrent arrhythmia for at least one year off all antiarrhythmic drugs, and confirmed by a cardiologist.
15. Have evidence or history of significant (controlled or uncontrolled) hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, renal, gastrointestinal, immunocompromising, or neurological disease, including seizure disorder, or any other medical disorder judged by the investigator to significantly increase the risk of MDMA administration (participants with hypothyroidism who are on adequate and stable thyroid replacement will not be excluded). Note: if participants present with a history of glaucoma, enrollment would be allowed only with the approval of their ophthalmologist
16. Have uncontrolled hypertension using the standard criteria of the American Heart Association (values of 140/90 milligrams of Mercury [mmHg] or higher assessed on three separate occasions)
17. Have a heart rate > 100 bpm on three separate occasions
18. Have a marked Baseline prolongation of QT/QTc interval (For purposes of eligibility, this is defined as repeated demonstration of a QT interval corrected using Fridericia's formula [QTcF] >450 milliseconds [ms] and >460 ms in females. For transgender or non-binary participants, QTc interval will be evaluated based on sex assigned at birth, unless the participant has been on hormonal treatment for five or more years.
19. Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
20. Require use of concomitant medications that prolong the QT/QTc interval during Experimental Sessions. Refer to Section 12.0 Concomitant Medications.
21. Have symptomatic liver disease
22. Have history of hyponatremia or hyperthermia
23. Are pregnant, nursing, or able to become pregnant and are not practicing an effective means of birth control.
24. Have hypersensitivity to any ingredient of the IMP (Investigational Medicinal Product).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of the intervention on Adjustment Disorder and relationship functioning in patients with cancer and a CSO. | 8 weeks ± 2 days
  The study will assess participants scores on The Adjustment Disorder New Module - 20 items (ADNM-20) from baseline to the primary time point (Visit 10, week 8 ± 2 days).
To assess the effectiveness of the intervention on Adjustment Disorder and relationship functioning in patients with cancer and a CSO. | 8 weeks ± 2 days
  The study will assess participants scores on the Couples Satisfaction Index (CSI-16) scores from baseline to the primary time point (Visit 10, week 8 ± 2 days).

SECONDARY OUTCOMES:
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 1) | 24 weeks
  Cancer patient: Edmonton Symptom Assessment System (ESAS)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 2) | 24 weeks
  Cancer Patient: Pain Interference Scale (PIS)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 3) | 24 weeks
  Cancer patient: Fatigue Assessment Scale (FAS)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 4) | 24 weeks
  Cancer patient: MAC scale
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 5) | 24 weeks
  Cancer patient and concerned significant other: Hospital Anxiety and Depression Scale (HADS A and D)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 6) | 24 weeks
  Cancer patient: Posttraumatic stress disorder CheckList-5 - Specific stressor (PCL-S)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 7) | 24 weeks
  Cancer patient and concerned significant other: Mystical Experience Questionnaire (MEQ)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 8) | 24 weeks
  Cancer patient and concerned significant other: Challenging Experience Questionnaire (CEQ)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 9) | 24 weeks
  Cancer patient: Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being 12 (FACIT-sp)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 10) | 24 weeks
  Cancer patient: Demoralization scale II (DS-II)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 11) | 24 weeks
  Cancer patient: Life Attitude Profile - revised, Death acceptance subscale (LAP-R; SAHD)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 12) | 24 weeks
  Cancer patient: Functional Assessment of Cancer Therapy - General (FACT-G)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 13) | 24 weeks
  Cancer patient: Family relationship Index (FRI)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 14) | 24 weeks
  Cancer patient and concerned significant other: Social Isolation Scale (SIS)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 15) | 24 weeks
  Cancer patient and concerned significant other: Everyday/illness-related disclosure (ELID)
To assess the effect on psychological distress, Mental Adjustment to Cancer (MAC), relationship functioning and health-related quality of life in both patients and their concerned significant other (scale 16) | 24 weeks
  Concerned significant other: CareGiver Oncology Quality of Life questionnaire (CarGOQoL)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Agrawal, MD, Principal Investigator — Sunstone Medical, PC
Locations (1):
- Sunstone Medical, PC, Rockville, Maryland, United States